CLINICAL TRIAL: NCT01682512
Title: Efficacy, Pharmacokinetics, and Safety of BI 695500 Versus Rituximab in Patients With Moderately to Severely Active Rheumatoid Arthritis: a Randomized, Double-blind, Parallel Arm, Multiple Dose, Active Comparator Trial.
Brief Title: Efficacy, Pharmacokinetics, and Safety of BI 695500 in Patients With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: substance discontinued
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1301.1; 2011-002894-48 (EudraCT Number)
Record Dates: First submitted 2012-08-10; First posted 2012-09-11 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

ARMS (5):
- Part I BI 695500 group (Experimental): BI 695500, Two infusions separated by 2 weeks, Intravenous infusion
  Interventions: Drug: BI 695500
- Part I Rituxan® (Active Comparator): rituximab, Two infusions separated by 2 weeks, Intravenous infusion
  Interventions: Drug: Rituxan®
- Part I MabThera® (Active Comparator): rituximab, Two infusions separated by 2 weeks, Intravenous infusion
  Interventions: Drug: MabThera®
- Part II BI 695500 group (Experimental): BI 695500, Two infusions separated by 2 weeks, Intravenous infusion
  Interventions: Drug: BI 695500
- Part II rituximab group (Active Comparator): rituximab, Two infusions separated by 2 weeks, Intravenous infusion
  Interventions: Drug: Rituxan®

INTERVENTIONS:
Drug: BI 695500
  Arms: Part II BI 695500 group
Drug: BI 695500
  Arms: Part I BI 695500 group
Drug: Rituxan®
  Arms: Part I Rituxan®
Drug: Rituxan®
  Arms: Part II rituximab group
Drug: MabThera®
  Arms: Part I MabThera®

SUMMARY:
The primary objectives of this trial are (1) To show PK (Pharmacokinetic) similarity of BI 695500 to rituximab. (2)To establish statistical equivalence of efficacy of BI 695500 and rituximab, in patients with moderately to severely active RA (Rheumatoid Arthritis), based on the change in Disease Activity Score 28 (DAS28) score measured at 24 weeks compared to Baseline and the American College of Rheumatology 20% (ACR20) response rate at Week 24.

ELIGIBILITY:
Inclusion criteria:

1. Must give written informed consent and be willing to follow the protocol.
2. Male or female participants, between 18 and 80 years of age, who have a diagnosis of moderately to severely active RA for at least 6 months as defined by at least six swollen joints (66 joint count) and at least eight tender joints (68 joint count) at Screening and Baseline (Day 1), and either an erythrocyte sedimentation rate (ESR) of > 28 mm/hour OR a C-reactive protein (CRP) level > 1.0 mg/dL (normal: < 0.4 mg/dL) at Screening. Patients must have had an inadequate response or intolerance to conventional DMARD therapy including at least one tumor necrosis factor (TNF) inhibitor.
3. Positive for Radio Frequency and/or anti-CCP (Anti-cyclic citrullinated peptide) antibodies.
4. Current treatment for RA on an outpatient basis:

   1. Must be currently receiving and tolerating oral or parenteral MTX therapy at a dose of 15-25 mg per week (dose may be as low as 10 mg per week if the patient is unable to tolerate a higher dose) for at least 12 weeks immediately prior to Day 1. The dose should be stable for at least 4 weeks prior to Day 1 until Week 24. After Week 24 the administration route can be changed at the investigator's discretion.
   2. Patients must be willing to receive oral folic acid (at least 5 mg/week or as per local practice) or equivalent during the entire study (mandatory co-medication for MTX treatment).
   3. Biologic agents and DMARDs (other than MTX) must be withdrawn at least 2 weeks prior to Day 1, except azathioprine and etanercept which must be withdrawn at least 4 weeks prior to Day 1; abatacept, adalimumab, anakinra, certolizumab, infliximab, and golimumab at least 8 weeks prior to Day 1; tocilizumab at least 10 weeks prior to Day 1.
   4. Leflunomide must be withdrawn at least 8 weeks prior to Day 1 or a minimum of 2 weeks prior to Day 1 if after 11 days of standard cholestyramine washout.
   5. If receiving current treatment with oral corticosteroids (other than intra-articular or parenteral), the dose must not exceed 10 mg/day prednisolone or equivalent. During the 4 weeks prior to Baseline (Day 1) the dose must remain stable.
   6. Intra-articular and parenteral corticosteroids are not permitted within 6 weeks prior to Baseline Day 1 or throughout the trial, with the exception of IV administration of 100 mg methylprednisolone 30 to 60 minutes prior to each infusion as this is part of the trial procedures.
   7. Any concomitant non-steroidal anti-inflammatory drugs (NSAIDs) must be stable for at least 2 weeks prior to Day 1.
   8. Patients may be taking oral hydroxychloroquine provided that the dose is not greater than 400 mg/day or chloroquine provided that the dose is not greater than 250 mg/day. These doses must have been stable for a minimum of 12 weeks prior to Day 1. The hydroxychloroquine or chloroquine treatment will need to be continued at a stable dose with the same formulation until the end of the trial.
5. For participants of reproductive potential (males and females), use of a reliable means of contraception (e.g., hormonal contraceptive, patch, intrauterine device, physical barrier) has to be used throughout trial participation. Females of child-bearing potential must also agree to use an acceptable method of contraception for 12 months following completion or discontinuation from the trial.

Exclusion criteria:

1. ACR functional Class IV or wheelchair/bed bound.
2. Primary or secondary immunodeficiency (history of, or currently active), including known history of human immunodeficiency virus infection.
3. History of positive purified protein derivative test (positive tuberculosis [TB] test) without treatment for TB infection or chemoprophylaxis for TB exposure.
4. Positive HIV or TB at screening.
5. Known coronary artery disease or significant cardiac arrhythmias or severe congestive heart failure (New York Heart Association classes III or IV), or interstitial lung disease observed on chest X-ray.
6. History of IgE-mediated (immunoglobulin E) or non-IgE-mediated hypersensitivity or known anaphylaxis to mouse proteins or a history of hypersensitivity to antibody therapy.
7. History of cancer including solid tumors, hematologic malignancies, and carcinoma in situ (except participants with previous resected and cured basal or squamous cell carcinoma, treated cervical dysplasia, or treated in situ Grade I cervical cancer within 5 years prior to the Screening Visit).
8. History of pancreatitis or current peptic ulcer disease.
9. Receipt of a live/attenuated vaccine within 12 weeks prior to the Screening Visit.
10. Any condition or treatment (including biologic therapies) that, in the opinion of the investigator, may place the patient at unacceptable risk during the trial.
11. Pregnancy or breast feeding.
12. History of, or current, inflammatory joint disease other than RA (e.g., gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease) or other systemic autoimmune disorder (e.g., systemic lupus erythematosus, inflammatory bowel disease, pulmonary fibrosis, or Feltys syndrome, scleroderma, inflammatory myopathy, mixed connective tissue disease, or any overlap syndrome).
13. Diagnosis of juvenile idiopathic arthritis, also known as juvenile RA, and/or RA before age 16.
14. Any surgical procedure, including bone/joint surgery/synovectomy (including joint fusion or replacement) within 12 weeks prior to the Screening Visit or planned within 24 weeks of the Screening Visit.
15. Lack of peripheral venous access.
16. Evidence of significant uncontrolled concomitant disease such as, but not limited to, nervous system, renal, hepatic, endocrine, or gastrointestinal disorders which, in the investigator's opinion, would preclude patient participation.
17. Known concurrent viral hepatitis or known positivity to HBe-ag, HBV DNA, HBV DNA polymerase, HCVRNA, anti HCV antibodies.
18. Known active infection of any kind (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization or treatment with IV anti-infectives within 4 weeks of the Screening Visit or completion of oral anti-infectives within 2 weeks of the Screening Visit.
19. History of deep space/tissue infection (e.g., fasciitis, abscess, osteomyelitis) within 52 weeks of the Screening Visit.
20. History of serious infection or opportunistic infection in the last 2 years.
21. Any neurological (congenital or acquired), vascular or systemic disorder that might affect any of the efficacy assessments, in particular, joint pain and swelling (e.g., Parkinson's disease, cerebral palsy, diabetic neuropathy).
22. Currently active alcohol or drug abuse or history of alcohol or drug abuse (as determined by the investigator) within 52 weeks of the Screening Visit.
23. Treatment with IV Gamma Globulin or the Prosorba® Column within 6 months of the Screening Visit.
24. Treatment with IV or intramuscular corticosteroids.
25. Previous treatment with a B cell modulating or cell depleting therapy.
26. Intolerance or contraindications to IV glucocorticoids.
27. AST (aspartate aminotransferase) or ALT (alanine aminotransferase)> 3 times ULN (Upper Limit of Normal)
28. Hemoglobin < 8.0 g/dL.
29. Levels of IgG < 5.0 g/L.
30. Absolute neutrophil count < 1500/µL.
31. Platelet count < 75000/µL.
32. Participation in any previous clinical trial within 12 weeks of Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2012-09-05 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2016-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (109):
- United States (53):
  - Rheumatology Associates, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Associates, P.C., Glendale, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Mesa, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - Medvin Clinical Research, Covina, California
  - TriWest Research Associates, LLC, El Cajon, California
  - Advanced Medical Research, LLC, Lakewood, California
  - Premiere Clinical Research, LLC, Lakewood, California
  - ProHealth Partners, Long Beach, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Arthritis Center Medical Group, Santa Maria, California
  - Westlake Medical Research, Thousand Oaks, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Nascimento, Joao (Private Practice), Bridgeport, Connecticut
  - Avail Clinical Research, LLC, DeLand, Florida
  - New Horizon Research Center, Miami, Florida
  - Arthritis Associates, Inc., Orlando, Florida
  - Family Clinical Trials, Incorporated, Pembroke Pines, Florida
  - Arthritis & Rheumatology Associates of Palm Beach, Tampa, Florida
  - Lovelace Scientific Resources, Incorporated, Venice, Florida
  - Coeur d'Alene Arthritis Clinical Trials, Coeur d'Alene, Idaho
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Apex Medical Research, Chicago, Illinois
  - International Clinical Research, Overland Park, Kansas
  - Columbia Medical Practice, PC, Columbia, Maryland
  - Klein and Associates, M.D., P.A., Cumberland, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - West Michigan Rheumatology, PLLC, Grand Rapids, Michigan
  - Arthritis Consultants, Inc, St Louis, Missouri
  - Westroads Clinical Research, Omaha, Nebraska
  - Summit Medical Group, Clifton, New Jersey
  - Atlantic Coast Research, Toms River, New Jersey
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - Arthritis and Osteoporosis Medical Associates, PLLC, Brooklyn, New York
  - Box Arthritis & Rheumatology of the Carolinas, Charlotte, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - STAT Research, Incorporated, Dayton, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, P.C., Duncansville, Pennsylvania
  - Office of Dr. Ramesh C. Gupta, Memphis, Tennessee
  - Center for Inflammatory Disease, Nashville, Tennessee
  - ClinRX Research LLC, Carrollton, Texas
  - Adriana Pop Moody Clinic PA, Corpus Christi, Texas
  - Heartland Research Associates, LLC, Houston, Texas
  - ClinRx Research LLC, McKinney, Texas
  - Heartland Research Associates, LLC, Webster, Texas
  - The Seattle Arthritis Clinic, PS, Seattle, Washington
  - Tacoma Center for Arthritis Research, PS, Tacoma, Washington
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
  - Mountain State Clinical Research, Clarksburg, West Virginia
- Argentina (7):
  - Instituto Médico CER, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Organización Médica de Investigación, Ciudad Autonoma Buenos Aires
  - APRILLUS, Ciudad Autonoma Buenos Aires
  - Instituto CAICI, Rosario
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
- AZ Groeninge - Campus Vercruysselaan, Kortrijk, Belgium
- Bulgaria (4):
  - MHAT - Kaspela, EOOD, Plovdiv
  - MHAT-Plovdiv AD, Plovdiv
  - MHAT Lyulin, Sofia
  - UMHAT, Clinic of Cardiology, Stara Zagora, Stara Zagora
- Aviva Medical Clinical Trials Group, Burlington, Ontario, Canada
- Chile (3):
  - Interin, Santiago
  - Centro Medico Prosalud, Santiago
  - Hospital Clínico Pontificia Universidad Católica de Chile, Santiago
- Germany (4):
  - Klinische Forschung Berlin-Buch GmbH, Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - SMO.MD GmbH, Magdeburg, Magdeburg
  - ZeFOR GmbH, Zerbst
- Greece (2):
  - Euroclinic of Athens, Athens
  - "Attikon" University General Hospital of Attica, Haidari
- Budai Irgalmasrendi Korhaz KHT., Budapest, Hungary
- St Vincent's University Hospital, Dublin, Ireland
- Mexico (4):
  - Hospital de Jesus, Cuauhtémoc
  - Hospital Universitario de Saltillo, Saltillo
  - Centro de Investigación del Noroeste, Tijuana
  - Clinical Research Institute, Tlanepantla
- Antonius Ziekenhuis, Sneek, Netherlands
- Poland (6):
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Wojewodzki Szpital Zespolony w Elblagu, Elblag
  - Specjalistyczny Osrodek Alergologiczno-Intern. ALL-MED, Krakow
  - Linea Corporis Chirurgia Plastyczna Sp. z o. o., Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw
- Portugal (6):
  - Hospital Garcia de Orta, EPE, Almada
  - Hospital Fernando Fonseca, EPE, Amadora
  - Centro Hospitalar do Baixo Vouga, E.P.E. Unidade de Aveiro, Aveiro
  - Instituto Português de Reumatologia, Lisbon
  - Centro Hospitalar do Porto, EPE, Porto
  - Hospital de Sao Teotónio, Viseu
- Spain (4):
  - Hospital A Coruña, A Coruña
  - Instituto Ferran de Reumatologia, Barcelona
  - Hospital Virgen Macarena, Seville
  - Hospital Nuestra Señora de Valme, Seville
- Ukraine (10):
  - CI of Healthcare Kharkiv CCH #8, Kharkiv, Kharkiv
  - Oleksandrivska Clinical Hospital, Kyiv
  - National Scientific Center Academician M.D. Strazhesko, Kyiv
  - Volyn Reg. Center of Cardiovascular Path. and Thrombolysis, Lutsk
  - Lviv Regional Clinical Hospital, Lviv, Lviv
  - M.V. Sklifosovskyi Poltava RCH, Poltava, Poltava
  - M.I. Pyrogov VRCH, Vinnytsia, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia, Vinnytsia
  - Vinnytsia M.I. Pyrogov NMU Ch of internal medicine #3, Vinnytsia
  - Zaporizhzhia Regional Clinical Hospital, Zaporizhzhia, Zaporizhzhia
- Whipps Cross University Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled into this multi-center, randomized, double-blind, parallel arm, multiple dose, active comparator 2 part trial from 27 September 2017. Trial was terminated on 3 September 2015 and last subject completed 28 October 2016.
Pre-assignment Details: 509 subjects were screened for eligibility to participate in the trial. 293 subjects met all inclusion and exclusion criteria and were randomised to receive treatment. 6 subjects were included in an open-label safety run-in prior to randomisation in Part-I.
Groups:
- BI 695500: Patients administered 1000 milligram per 100 milliliter (1000 mg per 100 mL) of BI 695500 concentrate for solution for intravenous (IV) infusion each at Day 1 and 15. Patients with response to treatment were administered additional infusions at Week 24 and 26.
- Rituxan®: Patients administered 1000 mg per 100 mL of Rituxan® injection for intravenous (IV) use each at Day 1 and 15. Patients with response to treatment were administered additional infusions at Week 24 and 26.
- MabThera®: Patients administered 1000 mg per 100 mL of MabThera® concentrate for solution for intravenous (IV) infusion each at Day 1 and 15. Patients with response to treatment were administered additional infusions at Week 24 and 26.
Period: Overall Study
Arm/Group | BI 695500 | Rituxan® | MabThera®
Started | 116 | 111 | 66
Randomized in Part-I | 66 | 65 | 66
Randomized in Part-II | 50 | 46 | 0
Completed | 44 | 40 | 48
Not Completed | 72 | 71 | 18
Not completed — Adverse Event | 6 | 5 | 2
Not completed — Withdrawal by Subject | 2 | 6 | 3
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Study terminated by sponsor | 46 | 43 | 0
Not completed — Lost to Follow-up | 3 | 0 | 2
Not completed — Protocol Violation | 2 | 3 | 2
Not completed — Primary lack of efficacy | 10 | 7 | 7
Not completed — Secondary lack of efficacy | 1 | 1 | 0
Not completed — Other than stated above | 2 | 4 | 2

BASELINE CHARACTERISTICS:
Population: The safety randomized analysis set (SAFR) contained all randomized subjects who received at least one dose of trial medication and subjects were classified according to treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 695500 | Rituxan® | MabThera® | Total
Number analyzed (Participants) | 116 | 110 | 65 | 291
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (10.46) | 54.0 (11.10) | 54.8 (12.22) | 54.5 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 96 | 52 | 242
  Male | 22 | 14 | 13 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change of Disease Activity Score 28 Erythrocyte Sedimentation Rate (DAS28 [ESR]) From Baseline to Week 24 (BI 695500 Versus Rituxan®) - Part I
Description: The DAS28 score was derived using the formula: DAS28 (ESR) = 0.56*√(TJC28) + 0.28*√(SJC28) + 0.70*ln(ESR) + 0.014*(GH), where, TJC28 = 28 joint count for tenderness, SJC28 = 28 joint count for swelling, Ln(ESR) = natural logarithm of ESR, GH = the General Health component of the DAS [score on a visual analogue scale (VAS) ranging from 0 (very well) to 100 (very poor)].
  DAS28 values range from 2.0 to 10.0 while higher values mean a higher disease activity. Low disease activity is defined as a DAS28 score of ≤ 3.2 and DAS28 remission is defined as a DAS28 score of < 2.6. A clinically important change in DAS28 score is defined as an improvement in DAS28 score of at least 1.2.
  The full analysis set (FAS) contained all randomized subjects who received at least one dose of trial medication, had at least one assessment of primary efficacy endpoint at Baseline and at post-baseline visit prior or at Week 24 visit.
Time Frame: Baseline and Week 24
Population: FAS. Since this endpoint was designed to establish statistical equivalence of efficacy of BI 695500 and Rituxan®, only subjects randomized to BI 695500 and Rituxan® in part-I of study are included.
Measure: Least Squares Mean (90% Confidence Interval); unit: Unit on scale
Arm/Group | BI 695500 | Rituxan®
Number analyzed (Participants) | 58 | 61
Unit on scale | -1.8 [-2.08 to -1.50] | -1.4 [-1.64 to -1.09]
Statistical Analysis 1: Comparison: BI 695500 vs Rituxan®; Test type: Non-Inferiority or Equivalence — Equivalence for the change in DAS28 (ESR) was evaluated based on the two-sided 90% Confidence Interval (CI) for the treatment difference with respect to the mean change in the DAS28(ESR) score compared to baseline. Null hypothesis of non-equivalence was to be rejected if the 90% CI is fully contained within the interval of [-0.5, 0.5]; Mixed Models Analysis — Model analyzed was: DAS28(ESR) change from Baseline at Week 24 = overall mean + treatment + DAS28(ESR) Baseline score + visit + visit by treatment interaction + baseline-by-visit interaction + random error; A restricted maximum likelihood (REML)-based Mixed-Effect Model Repeated Measure (MMRM) approach was used; Adjusted mean difference = -0.4, 90% CI 2-sided [-0.83 to -0.03] — Adjusted mean difference was calculated as: BI 695500 - Rituxan®

2. Primary Outcome: PK (Part I Only): AUC0-tz (Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration, Determined Over Both Dosages)
Description: Pharmacokinetic (PK) (Part I only): AUC0-tz (area under the plasma concentration versus time curve from time zero to the last measurable concentration, determined over both dosages). Time zero was the time the first dose started. Only subjects randomized in part I of this study are included. As per protocol all the following criteria had to be fulfilled for a patient to be defined as PK evaluable for the Pharmacokinetic analysis set (PKS):
  Full first and second dose given. Pre-dose concentration available prior to the second dose. Ability to estimate AUC during the infusion phases. Ability to estimate the AUC for the distribution phase after the second dose. Ability to estimate the terminal half-life (t1/2) after the second dose.
  gMean - Geometric Mean
Time Frame: Blood PK samples were collected at -00:05 (hours: min) prior to first infusion and 03:55, 24:00, 335:55, 338:00, 339:55, 342:00, 344:00, 360:00, 432:00, 504:00, 672:00, 1176:00, 1512:00, 2352:00 and 2688:00 after first infusion.
Population: Pharmacokinetic analysis set (PKS) consisted of all randomized subjects who were PK evaluable based on protocol defined criteria.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour(h)*Microgram(ug)/Milliliter (mL)
Arm/Group | BI 695500 | Rituxan® | MabThera®
Number analyzed (Participants) | 56 | 56 | 55
Hour(h)*Microgram(ug)/Milliliter (mL) | 171000 (41.1) | 167000 (40.5) | 193000 (37.9)
Statistical Analysis 1: Comparison: BI 695500 vs Rituxan®; The similarity of AUC(o- tz) was compared between treatment groups BI 695500 and Rituxan; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-tz)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 102.35, 90% CI 2-sided [90.50 to 115.76], Standard Error of Mean 107.700 — Adjusted ratio of gMeans: BI 695500 versus Rituxan®; standard error is geometric standard error
Statistical Analysis 2: Comparison: BI 695500 vs MabThera®; The similarity of AUC(o- tz) was compared between treatment groups BI 695500 and MabThera; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-tz)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 88.21, 90% CI 2-sided [78.24 to 99.46], Standard Error of Mean 107.500 — Adjusted ratio of gMeans: BI 695500 versus MabThera®; standard error is geometric standard error
Statistical Analysis 3: Comparison: Rituxan® vs MabThera®; The similarity of AUC(o- tz) was compared between treatment groups Rituxan and MabThera; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-tz)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 86.18, 90% CI 2-sided [76.50 to 97.09], Standard Error of Mean 107.449 — Adjusted ratio of gMeans: Rituxan® versus MabThera®; standard error is geometric standard error

3. Primary Outcome: PK (Part I Only): AUC0-inf Pred (Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity, Determined Over Both Dosages)
Description: PK (Part I only): AUC0-inf pred (area under the plasma concentration versus time curve from time zero to infinity, determined over both dosages, and extrapolated to infinity using predicted last observed quantifiable concentration). Time zero was the time the first dose started. Only subjects randomized in part I of this study are included.
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | BI 695500 | Rituxan® | MabThera®
Number analyzed (Participants) | 56 | 56 | 54
h*ug/mL | 174000 (42.2) | 169000 (42.0) | 202000 (35.3)
Statistical Analysis 1: Comparison: BI 695500 vs Rituxan®; The similarity of AUC(o-inf pred) was compared between treatment groups BI 695500 and Rituxan; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-inf pred)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 102.46, 90% CI 2-sided [90.26 to 116.30], Standard Error of Mean 107.939 — Adjusted ratio of gMeans: BI 695500 versus Rituxan®; standard error is geometric standard error
Statistical Analysis 2: Comparison: BI 695500 vs MabThera®; The similarity of AUC(o-inf pred) was compared between treatment groups BI 695500 and MabThera; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-inf pred)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 86.00, 90% CI 2-sided [76.38 to 96.82], Standard Error of Mean 107.404 — Adjusted ratio of gMeans: BI 695500 versus MabThera®; standard error is geometric standard error
Statistical Analysis 3: Comparison: Rituxan® vs MabThera®; The similarity of AUC(o-inf pred) was compared between treatment groups Rituxan and MabThera; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-inf pred)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 83.93, 90% CI 2-sided [74.57 to 94.47], Standard Error of Mean 107.386 — Adjusted ratio of gMeans: Rituxan® versus MabThera®; standard error is geometric standard error

4. Primary Outcome: PK (Part I Only): AUC0-336 (Area Under the Plasma Concentration Versus Time Curve From Time Zero to 336 Hours)
Description: PK (Part I only): AUC0-336 (area under the plasma concentration versus time curve from time zero to 336 hours after the first dose). Time zero was the time the first dose started. Only subjects randomized in part I of this study are included.
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | BI 695500 | Rituxan® | MabThera®
Number analyzed (Participants) | 56 | 56 | 55
h*ug/mL | 49800 (40.1) | 51900 (28.9) | 55600 (30.7)
Statistical Analysis 1: Comparison: BI 695500 vs Rituxan®; The similarity of AUC(0-336) was compared between treatment groups BI 695500 and Rituxan; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-336)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 95.87, 90% CI 2-sided [86.21 to 106.62], Standard Error of Mean 106.608 — Adjusted ratio of gMeans: BI 695500 versus Rituxan®; standard error is geometric standard error
Statistical Analysis 2: Comparison: BI 695500 vs MabThera®; The similarity of AUC(0-336) was compared between treatment groups BI 695500 and MabThera; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-336)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 89.46, 90% CI 2-sided [80.23 to 99.74], Standard Error of Mean 106.775 — Adjusted ratio of gMeans: BI 695500 versus MabThera®; standard error is geometric standard error
Statistical Analysis 3: Comparison: Rituxan® vs MabThera®; The similarity of AUC(0-336) was compared between treatment groups Rituxan and MabThera; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-336)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 93.31, 90% CI 2-sided [85.11 to 102.29], Standard Error of Mean 105.700 — Adjusted ratio of gMeans: Rituxan® versus MabThera®; standard error is geometric standard error

5. Primary Outcome: PK (Part I Only): Observed Cmax (Maximum Plasma Concentration, Determined After the Second Dose)
Description: PK (Part I only): observed Cmax (observed maximum plasma concentration, determined after the second dose). Only subjects randomized in part I of this study are included.
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (ug/mL)
Arm/Group | BI 695500 | Rituxan® | MabThera®
Number analyzed (Participants) | 56 | 56 | 55
microgram per milliliter (ug/mL) | 434 (31.1) | 462 (32.0) | 486 (28.1)
Statistical Analysis 1: Comparison: BI 695500 vs Rituxan®; The similarity of observed Cmax was compared between treatment groups BI 695500 and Rituxan; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(Cmax)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 93.97, 90% CI 2-sided [85.32 to 103.50], Standard Error of Mean 105.995 — Adjusted ratio of gMeans: BI 695500 versus Rituxan®; standard error is geometric standard error
Statistical Analysis 2: Comparison: BI 695500 vs MabThera®; The similarity of observed Cmax was compared between treatment groups BI 695500 and MabThera; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(Cmax)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 89.30, 90% CI 2-sided [81.51 to 97.83], Standard Error of Mean 105.657 — Adjusted ratio of gMeans: BI 695500 versus MabThera®; standard error is geometric standard error
Statistical Analysis 3: Comparison: Rituxan® vs MabThera®; The similarity of observed Cmax was compared between treatment groups Rituxan and MabThera; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(Cmax)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 95.02, 90% CI 2-sided [86.62 to 104.25], Standard Error of Mean 105.744 — Adjusted ratio of gMeans: Rituxan® versus MabThera®; standard error is geometric standard error

6. Secondary Outcome: Percentage of Patients Meeting the ACR20 (American College of Rheumatology 20% Response Criteria) at Week 24 in Both Part-I and II
Description: A subject has an ACR20 response if all of the following occur:
  * a > 20% improvement in the swollen joint count (66 joints)
  * a > 20% improvement in the tender joint count (68 joints)
  * a > 20% improvement in at least 3 of the following assessments: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, patient's assessment of physical function, as measured by the Health Assessment Questionnaire - Disability Index, or Acute phase reactant (C-reactive protein).
  The percentage of subjects meeting the ACR20 response criteria at Week 24 (part-I and II) is presented for subjects randomised to receive BI 695500, Rituxan and MabThera.
Time Frame: Week 24
Population: FAS. Missing data have been imputed according to LOCF (last observation carried forward) and/or NRI (Non Responder Imputation).
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695500 | Rituxan® | MabThera®
Number analyzed (Participants) | 94 | 90 | 64
Percentage of participants | 26.6 | 23.3 | 56.3

7. Secondary Outcome: PK (Part I Only): AUC0-inf, Ppk (Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity, Based on Individual Predicted Concentrations for Missing Data Derived From a Population PK Model, Determined Over Both Dosages)
Description: PK (Part I only): AUC0-inf, ppk. Time zero was the time the first dose started. Only subjects randomized in part I of this study are included. A modeling approach was used to impute missing values as well as impute missing concentrations after the first dose with a sampling schedule identical to the first 2 weeks after the second dose. A unit dose of 1000 mg was used in calculating the imputed values. The resulting dataset thus consisted of PK evaluable and PK non-evaluable patients with both measured as well as imputed concentration values. The prediction of these concentrations was based on a mixed effect modeling approach and included significant covariates as identified during the PK model development (including age, body surface area [BSA], body mass index [BMI], weight, gender, race, and formulation).
Time Frame: as for outcome 2
Population: Pharmacokinetic full analysis set (PKFS) included all randomized subjects with at least one valid PK concentration measurement. A valid PK concentration measurement is a value greater than lower limit of quantification as provided by Charles River.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | BI 695500 | Rituxan® | MabThera®
Number analyzed (Participants) | 66 | 65 | 65
h*ug/mL | 165000 (42.9) | 158000 (50.0) | 180000 (40.6)
Statistical Analysis 1: Comparison: BI 695500 vs Rituxan®; The similarity of AUC(0-inf, ppk) was compared between treatment groups BI 695500 and Rituxan; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-inf, ppk)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 104.49, 90% CI 2-sided [91.92 to 118.78], Standard Error of Mean 108.044 — Adjusted ratio of gMeans: BI 695500 versus Rituxan®; standard error is geometric standard error
Statistical Analysis 2: Comparison: BI 695500 vs MabThera®; The similarity of AUC(0-inf, ppk) was compared between treatment groups BI 695500 and MabThera; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-inf, ppk)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 91.39, 90% CI 2-sided [81.38 to 102.64], Standard Error of Mean 107.253 — Adjusted ratio of gMeans: BI 695500 versus MabThera®; standard error is geometric standard error
Statistical Analysis 3: Comparison: Rituxan® vs MabThera®; The similarity of AUC(0-inf, ppk) was compared between treatment groups Rituxan and MabThera; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on logarithmic scale: Ln(AUC0-inf, ppk)=overall mean+treatment effect+random error; Adjusted ratio of gMeans (%) = 87.47, 90% CI 2-sided [77.12 to 99.21], Standard Error of Mean 107.896 — Adjusted ratio of gMeans: Rituxan® versus MabThera®; standard error is geometric standard error

ADVERSE EVENTS:
Time Frame: From the first dose of study medication and prior to the last date of study medication plus 6 months (180 days); up to 48 weeks
Description: The safety randomized analysis set (SAFR) contained all randomized subjects who received at least one dose of trial medication and subjects were classified according to treatment received.
Arm/Group | BI 695500 | Rituxan® | MabThera®
Serious Adverse Events (participants affected / at risk) | 9/116 | 9/110 | 5/65
Other Adverse Events (participants affected / at risk) | 17/116 | 14/110 | 24/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695500 (N=116) | Rituxan® (N=110) | MabThera® (N=65)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 2 | 0
Anaphylactoid reaction (Immune system disorders) | 0 | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695500 (N=116) | Rituxan® (N=110) | MabThera® (N=65)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 5
Viral upper respiratory tract infection (Infections and infestations) | 8 | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Dizziness (Nervous system disorders) | 1 | 1 | 4
Headache (Nervous system disorders) | 5 | 7 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 4

LIMITATIONS AND CAVEATS:
The study program was terminated and this study was discontinued on 3 September 2015. As a result no patients receiving study treatment in Part II of the study reached Week 24, and no conclusions regarding the efficacy of BI 695500 can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.